CLINICAL TRIAL: NCT03483415
Title: Investigation of Analgesic Effect of Long Thoracic Nerve Blockade After VATS (Video-Assisted Thoracoscopic Surgery) Operation
Brief Title: Long Thoracic Nerve Blockade for Pain Treatment After Video-Assisted Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2018/02-01
Record Dates: First submitted 2018-03-19; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Nerve Block; Video-Assisted Thoracic Surgery
MeSH Terms: interventions — Morphine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, single-blind
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup L (Experimental): IV patient-controlled analgesia (PCA) morphine
  + Ultrasound guided Long thoracic nerve blockage with 5 ml % 0.25 bupivacaine
  Interventions: Drug: Morphine Sulfate; Drug: Bupivacaine
- Group P (Active Comparator): IV patient-controlled analgesia (PCA) morphine
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — Intravenous morphine infusion with PCA: Solution was concentration of 0.5 mg/mL. Loading dose of 1 mg, 0.5 mg of bolus dose and 20 min of locking time.
  Other Names: Morphine
Drug: Bupivacaine — Ultrasound guided Long thoracic nerve blockage with 5 ml % 0.25 bupivacaine
  Arms: Grup L

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) provides an opportunity to penetrate the thoracic cavity by video through an incision into the chest wall and facilitate surgical operation of lung pathologies.Various regional methods of anesthesia are currently being used to achieve this goal.

The aim of the study was to assess the effectiveness of Long thoracic nerve bloc on postoperative VATS analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class and underwent video-assisted thoracoscopic surgery (VATS).

Exclusion Criteria:

* Previous history of opioid use preoperatively,
* Allergy to local anesthetics,
* The presence of any systemic infection,
* Uncontrolled arterial hypertension,
* Uncontrolled diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | Postoperative 24 hours
  morphine consumption

SECONDARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0=no pain, 10=intolerable pain)
side effect (Hypotension) | Postoperative 24 hours
  side effect Hypotension
additional analgesic use | Postoperative 24 hours
  additional analgesic use
side effect (Nausea and vomiting) | Postoperative 24 hours
  Nausea and vomiting scale
  1. Nausea and vomiting scale (nausea-vomiting scale (NVS): 1. No nausea is present, 2. Mild nausea is present. 3. Severe nausea is present. 4. Vomiting is present) In case of a NVS score of >3, an anti-emetic drug was administered.
side effect (Ramsay Sedation Scale (RSS) | Postoperative 24 hours
  Ramsay Sedation Scale (Ramsay Sedation Scale (RSS) : 1. Anxiety, agitation are present; 2. Cooperated, awake; 3. Sedatized, response to commands; 4. Sleepy, immediately awoken by auditory stimulus or glabella tap; 5. Sleepy, deep response to auditory stimulus or glabella tap and 6. Sleepy, no response to auditory stimulus or glabella tap)

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, M.D, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital